CLINICAL TRIAL: NCT00603460
Title: A Phase-I/II Randomized Trial of Maintenance Vaccination Combined With Metronomic Cyclophosphamide w/wo Adoptive Transfer of CD3/CD28-CoStimulated T-Cells for Recurrent Ovarian or Primary Peritoneal Cancer Previously Vaccinated DCVax-L
Brief Title: DCVax-L Vaccination With CD3/CD28 Costimulated Autologous T-Cells for Recurrent Ovarian or Primary Peritoneal Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Northwest Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UPCC 01808
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cancer
Keywords: Ovarian Cancer; Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Cyclophosphamide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Biological: DCVax-L and T Cells
- B (Active Comparator)
  Interventions: Biological: DCVax-L and T Cells

INTERVENTIONS:
Biological: DCVax-L and T Cells — Arm A
  * Optional DCVax-L prior to chemotherapy
  * Apheresis
  * Chemotherapy for 3 days (IV fludarabine/cyclosphosphamide)
  * Infusion of activated T cells
  * DCVax-L vaccine
  * End of study visit
  Arm B
  * Optional DCVax-L prior to chemotherapy
  * Apheresis
  * Chemotherapy for 3 days (IV fludarabine/cyclosphosphamide)
  * Infusion of activated T cells
  * DCVax-L vaccine
  * Oral cyclophosphamide (one week on/one week off) for a total for a total of 6 weeks
  * End of study visit
  Other Names: Cytoxan; Avastin; DCVax-L

SUMMARY:
Subjects with recurrent epithelial ovarian carcinoma or primary peritoneal cancer, who have previously undergone vaccination in clinical study UPCC-11807 with DCVax-L, an autologous vaccine with DC loaded in vitro with autologous tumor lysate.

Phase I Subjects enrolled in this study will receive leukapheresis; followed by cyclophosphamide/fludarabine-induced lymphodepletion; followed by adoptive transfer of ex vivo CD3/CD28-costimulated vaccine-primed peripheral blood autologous T cells; followed by a single DCVax-L vaccination, to establish feasibility and safety of this approach.

Primary Objectives of Phase I

To determine the feasibility and safety of administering vaccine-primed, ex vivo CD3/CD28-costimulated autologous peripheral blood T cells in combination with DCVax-L vaccination, following lymphodepletion with high dose cyclophosphamide/fludarabine.

Phase II

Twenty-two additional subjects will be randomized to receive either:

* ARM-IIA: maintenance DCVax-L vaccination, in combination with oral metronomic cyclophosphamide, or
* ARM-IIB: leukapheresis, followed by cyclophosphamide/fludarabine-induced lymphodepletion, followed by adoptive transfer of ex vivo CD3/CD28-costimulated vaccine-primed peripheral blood autologous T cells, followed by maintenance DCVax-L vaccination, plus oral metronomic cyclophosphamide.

Primary Objective of Phase II

To assess the distribution of progression-free survival at 6 months for patients treated with maintenance DCVax-L vaccination plus oral metronomic cyclophosphamide as well as patients treated with ex vivo CD3/CD28-costimulated vaccine-primed peripheral blood autologous T cells after lymphodepletion with high dose cyclophosphamide / fludarabine, followed by DCVax-L boost vaccination and metronomic oral cyclophosphamide.

DETAILED DESCRIPTION:
Description of treatment for Phase I:

* Patients will be offered, if medically indicated, tumor resection or needle aspiration of malignant effusion in order to make additional doses of DCVax-L vaccine.
* If subjects have not received DCVax-L vaccination within the last 3-4 weeks, and if DCVax-L is available, subjects have the option of receiving one dose of DCVax-L after enrolment, to boost the frequency of vaccine-primed T cells.
* Subjects will receive a single course of outpatient lymphodepleting chemotherapy with intravenous cyclophosphamide (300 mg/m2/d for 3 days) and intravenous fludarabine (30 mg/m2/d for 3 days) both administered on days 8 to 10.
* Ex vivo CD3/CD28-costimulated lymphocytes will be infused ~2 days after last day of fludarabine infusion.
* Patients will receive DCVax-L vaccine ~24-48 hrs after T cell infusion.
* Subjects will be contacted every 6 months for 5 years for survival.

Description of treatment for Phase II:

In ARM-IIA:

* Patients will be offered, if medically indicated, tumor resection or needle aspiration of malignant effusion in order to make additional doses of DCVax-L vaccine.
* Subjects will receive intradermal vaccinations with DCVax-L every 8 weeks, for four cycles total. The first vaccine will be administered on day 0, which can be no sooner than 4 weeks from previous DCVax-L vaccination related to clinical study UPCC-11807.
* Subjects will receive oral cyclophosphamide at metronomic schedule and dose (50 mg daily) every other week, starting ~3 weeks after DCVax-L in every vaccine cycle.
* Patients will be offered (with the right to refuse) CT-guided needle biopsy or needle aspiration of malignant effusion after the second vaccine.

In ARM-IIB:

* Patients will be offered, if medically indicated, tumor resection or needle aspiration of malignant effusion in order to make additional doses of DCVax-L vaccine.
* Subjects will undergo ~10-15 liter leukapheresis to derive vaccine-primed peripheral blood lymphocytes (PBL) on day 0. The apheresis material will be transferred to the Cell and Vaccine Facility at the University of Pennsylvania (Penn CVPF) for T cell manufacturing.
* If subjects have not received DCVax-L vaccination within the last 3-4 weeks, and if DCVax-L is available, subjects have the option of receiving one dose of DCVax-L after enrolment, to boost the frequency of vaccine-primed T cells.
* Subjects will receive a single course of outpatient lymphodepleting chemotherapy with intravenous cyclophosphamide (300 mg/m2/d for 3 days) and intravenous fludarabine (30 mg/m2/d for 3 days).
* Ex vivo CD3/CD28-costimulated lymphocytes will be infused ~2 days after last day of fludarabine infusion.
* Patients will receive DCVax-L vaccine boosts every 8 weeks for a total of four vaccines. The first DCVax-L will be given ~24-48 hrs after T cell infusion.
* Following DCVax-L, subjects will receive oral cyclophosphamide at metronomic schedule and dose (50 mg daily) every other week x 3 cycles, starting ~3 weeks after DCVax-L in every vaccine cycle.
* Patients will be offered (with the right to refuse) CT-guided needle biopsy or needle aspiration of malignant effusion ~1-2 weeks after the second vaccine

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in UPCC 11807 (A Phase I Clinical Trial of Autologous Dendritic Cell Vaccine Loaded with Autologous Tumor Cell Lysate for Recurrent Ovarian or Primary Peritoneal Cancer)
* PS < 2
* Subject must have tumor lysate sufficient to prepare at least 4 DCVax-L vaccines
* 18 years of age or older
* Life expectancy > 4 months
* Signed Informed Consent
* Normal organ and bone marrow function defined by:
* ANC ≥ 1,000/μl
* Platelets >100,000/μl
* AST(SGOT)/ALT(SGPT) < 2.5 X institutional upper limit of normal
* Bilirubin <2.0 mg/dL unless secondary to bile duct blockage by tumor
* Creatinine <1.5 X the upper limit of normal

Exclusion Criteria:

* Subjects with the following:
* known brain metastases
* renal insufficiency
* liver failure
* organ allograft
* known autoimmune/collagen vascular disorders
* pregnant or breast feeding
* non-healing wounds, ulcers, or bone fractures
* positive for serum anti-Yo (cdr2) antibodies
* uncontrolled hypertension
* Myocardial infarction or unstable angina within 6 months prior to registration
* New York Heart Association (NYHA) Grade II or greater congestive heart failure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Disease status will be assessed with CT (or MRI) of chest/abdomen/pelvis at enrollment, after vaccine 2 and at the conclusion of the study . Rates of disease progression will be recorded at the time of study conclusion. | Enrollment, 3 months after enrollment, End of study

CONTACTS AND LOCATIONS:
Overall Officials: George Coukos, M.D., Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylania, Philadelphia, Pennsylvania, United States